CLINICAL TRIAL: NCT07168850
Title: Focused Ultrasound Pallidotomy for Medication-Refractory Limb Dystonia (FUTURE Study)
Brief Title: Focused Ultrasound Unilateral Pallidotomy for Medication-Refractory Limb Dystonia
Acronym: FUTURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: Azienda ULSS 3 Serenissima (Other); IRCCS Centro Neurolesi Bonino Pulejo (Other); Azienda Ospedaliera Villa Sofia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PNRR-MCNT2-2023-12378417
Record Dates: First submitted 2025-08-20; First posted 2025-09-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-09

CONDITIONS: Limb Dystonia; Idiopathic Dystonia; Medication-refractory Dystonia; Dystonia, Focal
Keywords: Focused Ultrasound; MRgFUS; Pallidotomy; Dystonia; Exablate; Neuromodulation; fMRI; TMS
MeSH Terms: conditions — Dystonia; Dystonic Disorders

STUDY DESIGN:
Intervention Model Description: 34 adult patients (17 per arm) will be randomized to receive either active MRgFUS pallidotomy or a sham procedure. Patients in the sham group will cross over to active treatment at 3 months. The follow-up period for all patients will be 6 months post-treatment.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double-blind (Participant, Care Provider, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Pallidotomy (MRgFUS) (Experimental): Patients undergo unilateral pallidotomy using Exablate system under MRI guidance.
  Interventions: Device: Exablate MR-guided Focused Ultrasound Pallidotomy
- Sham Procedure (Sham Comparator): Identical setup without thermal lesioning. Participants cross over to active Pallidotomy after 3 months.
  Interventions: Device: Exablate MR-guided Focused Ultrasound Pallidotomy; Device: Sham Sham Exablate MRgFUS Pallidotomy

INTERVENTIONS:
Device: Exablate MR-guided Focused Ultrasound Pallidotomy — Active Pallidotomy
Device: Sham Sham Exablate MRgFUS Pallidotomy — Sham procedure. Identical setup without thermal lesioning. Participants cross over to Active Pallidotomy after 3 months.
  Arms: Sham Procedure

SUMMARY:
The goal of this clinical trial is to find out if a non-invasive procedure called focused ultrasound can safely and effectively treat limb dystonia in adults who have not improved with medications or botulinum toxin injections.

The main questions it aims to answer are:

* Does focused ultrasound reduce the severity of limb dystonia symptoms?
* Is the procedure safe and well tolerated?

Researchers will compare people who receive focused ultrasound treatment to those who receive a sham procedure (a look-alike procedure without active treatment) to see if the treatment works.

Focused ultrasound works by producing a very small (millimeter-size) lesion in a deep brain region. In this study, the lesion is located in a region called globus pallidus, which helps control movement.

Participants will:

* Be randomly assigned to one of two groups: focused ultrasound or sham
* Undergo a procedure using MRI and focused ultrasound to target a part of the brain called the globus pallidus
* Be followed for 6 months after treatment to assess changes in symptoms, quality of life, and brain function
* Participants in the sham group will be offered the real treatment after 3 months

This study may offer a new non-surgical treatment option for people with dystonia affecting the arm or leg, whose pharmacological control is unsatisfactory.

DETAILED DESCRIPTION:
The FUTURE study is a prospective, randomized, double-blind, sham-controlled, multicenter national clinical trial aimed at assessing the efficacy and safety of unilateral MR-guided focused ultrasound (MRgFUS) pallidotomy in patients with limb dystonia that is refractory to standard pharmacological treatments.

Dystonia is a movement disorder characterized by sustained or intermittent muscle contractions, causing abnormal movements or postures. In many cases, focal or segmental dystonias affecting the limbs can be managed with oral medications and botulinum toxin (BoNT) injections. However, a subset of patients does not respond adequately to these treatments. For such individuals, surgical intervention may offer relief, yet it remains underutilized due to concerns about invasiveness and complications.

Recent advancements in non-invasive neurosurgical techniques have introduced MRgFUS pallidotomy, a procedure that uses focused ultrasound beams under real-time MRI guidance to precisely ablate small brain targets-in this case, the globus pallidus internus (GPi). The FUTURE study specifically explores this technique as a less invasive alternative to deep brain stimulation, especially for patients with focal or segmental limb dystonia who are ineligible or reluctant to undergo conventional surgery.

The trial will enroll 34 adult patients with idiopathic or genetic limb dystonia that has proven resistant to pharmacologic and BoNT treatment. These patients will be randomly assigned in a 1:1 ratio to either:

* an active treatment group, undergoing unilateral GPi lesioning via MRgFUS,
* or a sham control group, receiving the same procedural setup but without therapeutic sonications.

At three months post-randomization, all patients in the sham group will cross over to receive the active MRgFUS treatment, allowing within-subject comparisons while ensuring ethical access to the therapeutic intervention. The follow-up period for each patient will last six months after active treatment, totaling a maximum of nine months of participation.

The primary endpoint is the change in motor severity as measured by the Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) at three months post-treatment. Secondary endpoints include adverse event frequency, patient and clinician global impressions of change, disability assessments (e.g., QuickDASH), quality of life (SF-36), and neurocognitive testing.

Additionally, the study will incorporate neurophysiological (TMS) and neuroimaging (resting-state fMRI) techniques to investigate treatment-induced changes in cortical excitability, plasticity, and functional connectivity, providing insight into the neural mechanisms underlying clinical improvement.

The FUTURE study is coordinated by the Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy with participation from other three major Italian neurological institutes. It represents a pioneering effort to evaluate focused ultrasound as a non-invasive therapeutic option for patients with disabling and treatment-resistant forms of limb dystonia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Able and willing to consent and attend visits
* Idiopathic or hereditary limb dystonia (focal, segmental, or multifocal; isolated or combined)
* Refractory to oral therapy and botulinum toxin
* Stable medication for ≥30 days and ≥90 days since last BoNT
* Capable of communicating during Exablate procedure

Exclusion Criteria:

* Acquired secondary dystonia
* Dementia or other neurodegenerative disorders
* Any clinically significant or unstable medical condition, which, in the opinion of the principal investigator or the clinician delegated by the principal investigator, may put the participant at risk when participating in the study (e.g., unstable heart disease or coagulopathy; uncontrolled psychiatric comorbidity)
* Prior deep brain stimulation or other brain surgery
* Any contraindication to MRI
* Skull Density Ratio (SDR) < 0.40
* Significant brain lesions (eg brain tumor, significant white matter lesions or globus pallidus interna lesions on baseline MRI)
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Chenge in the Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) | Baseline to Week 12
  The BFMDRS has a maximum score of 120 for the movement subscale and 30 for the disability subscale. Higher scores indicating more severe dystonia.

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events | Baseline to Week 24
  Assessment of any treatment-related adverse events throughout the whole study period
Changes in the Quick Disabilities of Arm, Shoulder & Hand (Quick-DASH) score | Baseline, Week 12 and Week 24
  The QuickDASH is a shortened, 11-item version of the DASH Outcome Measure, designed to assess physical function and symptom severity related to the arm, shoulder, and hand. Maximum score 100; the greater the score the grear the disability.
Changes in the Clinical Global Impression of Change (CGIC) score | Baseline, week 12 and week 24
  The CGIC is a 7-point scale used to assess the degree of change in a patient's condition since the start of treatment or another defined baseline. Lower scores indicates improvement and higher scores indicating worsening of the patient's condition.
Patient Global Impression of Change (PGIC) | Baseline, Week 12 and week 24
  The maximum score of the PGIC is 7: the higher the score the higher the improvement reported by a patient.
Change in the 36-Item Short Form Survey (SF-36) score | Baseline, week 12 and week 24
  The SF-36 questionnaire has a maximum score of 100 for each of its eight scaled scores (physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health). The higher the scores the more favorable is health state within that specific dimension.
Changes in the Short-Interval Cortical Inhibition (SICI) | Baseline and Week 24
  This is a neurophysiological measure of inhibitory processes within the motor cortex, assessed using Transcranial Magnetic Stimulation, which is measured as the relative amplitude reduction of motor evoked potentials from the test stimulus when it is preceded by the conditioning stimulus. The greater the change in SICI, the greater the pallidotomy-induced changes in motor cortex intracortical inhibitory circuits
Changes in intracortical facilitation (ICF) | Baseline and Week 24
  This is a neurophysiological measures of cortical excitability, assessed using paired-pulse Transcranial Magnetic Stimulation, which describes an increase in the magnitude of a motor evoked potential in a target muscle when a suprathreshold test pulse is preceded by a subthreshold conditioning pulse at specific interstimulus intervals. The greater the change in ICF, the greater the pallidotomy-induced changes in intracortical excitatory circuits
Changes in Paired Associative Stimulation (PAS) | Baseline and week 24
  This is a neurophysiological measure of cortical plasticity assessed using transcranial magnetic stimulation. The greater the change in PAS, the greater the pallidotomy-induced changes in motor cortex synaptic plasticity
Changes in brain activity (using functional connectivity) using resting-state functional magnetic resonance imaging (rs-fMRI) | Baseline and Week 24
  The investigators will conduct a region-of-interest analysis to calculate changes of fMRI functional connectivity between baseline and post-pallidotomy.
Changes in pallidotomy lesion morphology via contrast MRI | 24-hour after the procedure, week 12 and week 24
  To evaluate the morphological changes of the lesion after 24 hours, 3 months and 6 months from pallidotomy using contrast-enhanced brain MRI and their relationship with clinical changes including adverse events.
Changes in the Montreal Cognitive Assessment (MoCA) score | Baseline, week 12 and week 24
  Changes in the Montreal Cognitive Assessment (MoCA) score, a 30-point test of global cognitive functions. Score range: 0-30, with lower scores indicating worse cognitive function and higher scores indicating better cognitive function.
Change in Digit Span test score | Baseline, week 12 and week 24]
  Change in Digit Span test score, a cognitive test assessing memory functions. Score range: 0-[insert maximum score for the test], with lower scores indicating greater memory impairment and higher scores indicating better memory function.
Change in the Stroop Test score | Baseline, week 12 and week 24
  Change in Stroop Test scores, a neuropsychological test assessing frontal-lobe executive cognitive function. Score range: [insert minimum]-[insert maximum], with higher scores or slower reaction times indicating worse executive cognitive function.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Azienda ULSS3 Serenissima, Mestre, (Venice)
  - IRCCS Centro Neurolesi "Bonino-Pulejo", Messina
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia, Palermo

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request with appropriate safeguards for privacy and confidentiality
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement. For more information or to submit a request, please contact the P.I. of the study

REFERENCES:
- [Background] Rothwell JC, Hallett M, Berardelli A, Eisen A, Rossini P, Paulus W. Magnetic stimulation: motor evoked potentials. The International Federation of Clinical Neurophysiology. Electroencephalogr Clin Neurophysiol Suppl. 1999;52:97-103. No abstract available. PMID 10590980
- [Background] Sohn YH, Hallett M. Disturbed surround inhibition in focal hand dystonia. Ann Neurol. 2004 Oct;56(4):595-9. doi: 10.1002/ana.20270. PMID 15455393
- [Background] Burke RE, Fahn S, Marsden CD, Bressman SB, Moskowitz C, Friedman J. Validity and reliability of a rating scale for the primary torsion dystonias. Neurology. 1985 Jan;35(1):73-7. doi: 10.1212/wnl.35.1.73. PMID 3966004
- [Background] Horisawa S, Yamaguchi T, Abe K, Hori H, Fukui A, Iijima M, Sumi M, Hodotsuka K, Konishi Y, Kawamata T, Taira T. Magnetic Resonance-Guided Focused Ultrasound Thalamotomy for Focal Hand Dystonia: A Pilot Study. Mov Disord. 2021 Aug;36(8):1955-1959. doi: 10.1002/mds.28613. Epub 2021 May 29. PMID 34050695
- [Background] Stieglitz LH, Mahendran S, Oertel MF, Baumann CR. Bilateral Focused Ultrasound Pallidotomy for Parkinson-Related Facial Dyskinesia-A Case Report. Mov Disord Clin Pract. 2022 May 9;9(5):647-651. doi: 10.1002/mdc3.13462. eCollection 2022 Jul. PMID 35844284
- [Background] Krishna V, Fishman PS, Eisenberg HM, Kaplitt M, Baltuch G, Chang JW, Chang WC, Martinez Fernandez R, Del Alamo M, Halpern CH, Ghanouni P, Eleopra R, Cosgrove R, Guridi J, Gwinn R, Khemani P, Lozano AM, McDannold N, Fasano A, Constantinescu M, Schlesinger I, Dalvi A, Elias WJ. Trial of Globus Pallidus Focused Ultrasound Ablation in Parkinson's Disease. N Engl J Med. 2023 Feb 23;388(8):683-693. doi: 10.1056/NEJMoa2202721. PMID 36812432
- [Background] Hariz M. Pros and Cons of Ablation for Functional Neurosurgery in the Neurostimulation Age. Neurosurg Clin N Am. 2023 Apr;34(2):291-299. doi: 10.1016/j.nec.2022.11.006. Epub 2023 Jan 30. PMID 36906335
- [Background] Horisawa S, Fukui A, Takeda N, Kawamata T, Taira T. Safety and efficacy of unilateral and bilateral pallidotomy for primary dystonia. Ann Clin Transl Neurol. 2021 Apr;8(4):857-865. doi: 10.1002/acn3.51333. Epub 2021 Mar 15. PMID 33720521
- [Background] Centen LM, Oterdoom DLM, Tijssen MAJ, Lesman-Leegte I, van Egmond ME, van Dijk JMC. Bilateral Pallidotomy for Dystonia: A Systematic Review. Mov Disord. 2021 Mar;36(3):547-557. doi: 10.1002/mds.28384. Epub 2020 Nov 20. PMID 33215750
- [Background] Jankovic J. Medical treatment of dystonia. Mov Disord. 2013 Jun 15;28(7):1001-12. doi: 10.1002/mds.25552. PMID 23893456
- [Background] Hallett M, Benecke R, Blitzer A, Comella CL. Treatment of focal dystonias with botulinum neurotoxin. Toxicon. 2009 Oct;54(5):628-33. doi: 10.1016/j.toxicon.2008.12.008. Epub 2008 Dec 13. PMID 19103214